CLINICAL TRIAL: NCT04987632
Title: Effect of Acupuncture Plus Governor Vessel Moxibustion Combined With Letrozole on Live Birth in Anovulatory Infertile Women With Spleen-kidney Yang Deficiency Polycystic Ovary Syndrome: a Randomised Controlled Trial
Brief Title: Effect of Acupuncture Plus Governor Vessel Moxibustion Combined With Letrozole on Live Birth in Anovulatory Infertile Women With Spleen-kidney Yang Deficiency PCOS
Acronym: PCOS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qiu-ping Lin (Other)
Responsible Party: Sponsor-Investigator, Qiu-ping Lin, Sponsor-Investigator, Dongguan Hospital of Traditional Chinese Medicine
Organization: Dongguan Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20211408
Record Dates: First submitted 2021-07-15; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: PCOS; Infertility, Female
Keywords: PCOS; acupuncture; Governor vessel moxibustion; spleen-kidney Yang deficiency; letrozole
MeSH Terms: conditions — Infertility, Female | interventions — Letrozole; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letrozole combined with acupuncture and Du Meridian moxibustion group (Experimental): Letrozole combined with acupuncture and Du Meridian moxibustion was taken from 3-5 days of menstrual period (spontaneous menstruation or progesterone withdrawal bleeding). The acupuncture treatment was 3 times / week, with an interval of 2-4 days, 12 times a week, 30 minutes each time; Du Meridian moxibustion is 20 minutes each time, once a week, four times a week. The initial dose of letrozole was 2.5mg/day for 5 consecutive days. The follow-up dose was determined according to the response of the subjects to the initial dose, with one month as a cycle. If not pregnant, the subjects received letrozole for up to 4 cycles to induce ovulation with acupuncture plus Du Meridian moxibustion.
  Interventions: Drug: Letrozole; Device: acupuncture; Other: Governor vessel moxibustion
- Letrozole group (Active Comparator): Letrozole was taken 3-5 days after menstruation (spontaneous menstruation or progesterone withdrawal bleeding). The initial dose of letrozole was 2.5mg/day for 5 consecutive days. The follow-up dose was determined according to the response of the subjects to the initial dose, with one month as a cycle. In the absence of pregnancy, subjects were treated with letrozole for up to four cycles.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Letrozole, an aromatase inhibitor, is considered to be the first-line drug for ovulation induction in PCOS.
Device: acupuncture — Domestic and foreign studies suggest that acupuncture and electroacupuncture can improve the menstrual cycle of PCOS and reduce the level of total testosterone; Acupuncture can regulate glucose homeostasis by stimulating the autonomic nervous system of PCOS patients. Our previous studies and a large number of literatures have proved that acupuncture can improve insulin resistance in PCOS, and acupuncture can improve the pregnancy rate in PCOS.
  Arms: Letrozole combined with acupuncture and Du Meridian moxibustion group
Other: Governor vessel moxibustion — It can warm the kidney, promote digestion and absorption, remove dampness and promote blood circulation
  Arms: Letrozole combined with acupuncture and Du Meridian moxibustion group

SUMMARY:
Investigators expected to verify this hypothesis through this study:acupuncture and moxibustion combined with LE induced ovulation in Chinese anovulatory PCOS women has a higher rate of live birth than LE induced ovulation alone.

DETAILED DESCRIPTION:
It is a prospective, single center, clinical, randomized, controlled study. The subjects were 90 PCOS anovulatory participants of spleen kidney yang deficiency type, aged 20-40 years, who were treated in the outpatient department of Obstetrics and Gynecology of Dongguan Hospital of traditional Chinese medicine from January 2021 to December 2022. Participants were randomly divided into two groups: Acupuncture plus Du Meridian moxibustion combined with LE ovulation induction treatment group and single Le ovulation induction control group, 45 cases in each group.

The subjects in the two groups began to take letrozole or combined with acupuncture and Du Meridian moxibustion on 3-5 days of menstruation (spontaneous menstruation or progesterone withdrawal bleeding). If not pregnant, the subjects received letrozole for up to 4 cycles to induce ovulation or acupuncture plus Du Meridian moxibustion. Once pregnancy is found, acupuncture and Du Meridian moxibustion or drug treatment will stop immediately.

At the end of treatment, data were collected to observe the differences of live birth rate, pregnancy rate, ovulation rate, sex hormone, steroid hormone, glucose and lipid metabolism index and safety index between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 20 and 40.
* It meets the diagnostic criteria of spleen-kidney Yang deficiency type PCOS.
* According to World Health Organization standards (2010), the husband's semen analysis meets ① or ②.①Sperm density ≥15×10^6/ml, and motile sperm (forward and non-forward) ≥40% (A + B + C ≥40%)).② Total motile sperm number ≥9 million.That is, the percentage of semen volume × semen density × motility sperm ≥9×10^6.
* Tubal patency tests, including hysterosalpingography and diagnostic laparoscopy, which show that at least one fallopian tube is open.(If there is no history of pelvic operation or abortion, patency test results are effective within 3 years;If there is a history of fertility within 5 years and there is no pelvic operation, the tubal patency test is not required).
* Agree to discontinue the use of other therapies during the study. 6) Participate in the study voluntarily and sign the informed consent.

Exclusion Criteria:

* Eliminate other endocrine disorders: ① Patients with hyperprolactinemia (defined as two prolactin levels greater than or equal to 25ng/ml or determined by local standard values at least one week apart).The goal of excluding patients with hyperprolactinemia was to reduce variability among PCOS patients.These patients may be treated with alternative therapies (e.g., dopamine agonists).Those who had received treatment within the past year or were receiving treatment with normal test values could be enrolled. ② Menopausal FSH level (> 15 mIU/mL).Normal levels in the past year are eligible for inclusion. ③ Patients with uncorrected thyroid disease (defined as TSH < 0.2 mIU/mL or >5.5 mIU/mL).In the past year, normal levels can be included in the group. ④ Patients with poorly controlled type I or II diabetes (defined as a bb0 7.0% glycosylated hemoglobin level) or patients receiving antidiabetic drugs such as insulin, thiazole-lowering drugs, acarbose, or sulfonylureas may obfuscate the effects of the study drugs;Patients who were being treated with metformin in order to be diagnosed with type I or II diabetes or PCOS also need to be excluded. ⑤ Suspected patients with Cushing syndrome.
* In the last 2 months, use of hormones or other drugs, including TCM prescriptions and Chinese patent medicines, may affect the results.
* Pregnancy history within the last 6 weeks.
* A history of miscarriage or birth in the last 6 weeks.
* A history of breastfeeding in the last 6 months.
* Do not agree to sign the informed consent for this study.
* PCOS women who do not belong to the syndrome of spleen-kidney Yang deficiency.
* Special exclusion criteria： ① Patients with adrenal or ovarian tumors suspected of producing androgens. ② Both the husband and wife have had sterilization operations (vasectomy, tubal ligation) before, and the ligation has been loosened.Previous surgery may have influenced the results of the study.Patients with both husband and wife having undergone sterilization and PCOS at the same time are rare, and the inclusion of these patients should be excluded, otherwise the progress of this study will be affected. ③ Patients who have had bariatric surgery recently (<12 months) and who are in a period of dramatic weight loss or who have had bariatric surgery to prohibit pregnancy. ④ Untreated hypertensive patients with poor blood pressure control were defined as ≥60min between two blood pressure measurements, ≥160 mm Hg systolic or ≥100 mm Hg diastolic. ⑤ Patients with known congenital adrenocortical hyperplasia. ⑥ Oral ontraceptives, progesterone or hormone implants (including subcutaneous implants).A 2-month clearance period is required before screening of patients who have received these drugs.Storage of contraceptive forms or implants, especially if the implants have not been removed, may require longer removal time.Oral contraceptives take about a month to clear the drug. ⑦ Patients with liver disease with AST or ALT >2 times normal value or total bilirubin >2.5 g/dL.Patients with nephropathy with BUN > 30 mg/dL or serum creatinine > 1.4 mg/dL. ⑧ Patients with significant anemia (hemoglobin < 10 g/dL). ⑨Patients with a history of deep vein thrombosis, pulmonary embolism, or cerebrovascular disease .⑩ Patients with heart disease that may worsen after pregnancy. ⑪ Patients with a suspected history of cervical, endometrial or breast cancer.Women 21 years of age and older should have normal results from a Pap smear or TCT test. ⑫ Patients with a current history of alcoholism.Binge drinking was defined as > 14 times a week or binge drinking. ⑬ Patients also participated in other clinical studies.These studies require medication, sex restriction, or other barriers to compliance. ⑭ Patients who are expected to discontinue treatment for more than 1 month during the study period should not be included. ⑮ Patients taking other medications known to affect reproductive function or metabolism.These drugs include oral contraceptives, GnRH agonists and antagonists, antiandrogens, gonadotropins, anti-obesity drugs, anti-diabetic drugs such as metformin and thiazolidindiones, growth hormone release inhibiting hormones, diazazines, ACE inhibitors, and calcium channel blockers.The removal time of the above drugs should be 2 months.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-08-03 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
live birth rate | Within 1 year after the end of Cycle 4 (each cycle is 28 days).
  Ratio of the number ofdelivery of a live-born infant to the total number pregnancies of trials.
Clinical pregnancy rate | From the beginning to 14 days after the end of cycle 4 (each cycle is 28 days).
  Ratio of the number of pregnancies to the total number of trials.

SECONDARY OUTCOMES:
Ovulation rate | From the beginning to 14 days after the end of cycle 4 (each cycle is 28 days).
  Ratio of total ovulation times to the sum of the number of trials in each cycle(each cycle is 28 days).
Multiple pregnancy rate | From the beginning to 14 days after the end of cycle 4 (each cycle is 28 days).
  The rate of multiple pregnancies to total pregnancies.
Abortion rate | From the beginning to 14 days after the end of cycle 4 (each cycle is 28 days).
  Ratio of miscarriage in the total number of pregnancies.
HOMA-IR | Before the trail and at the end of cycle 4.
  Insulin resistance index is equal to fasting blood glucose multiplied by fasting insulin ratio 22.5. Recently, it was proposed that insulin resistance should be judged when it is greater than 2.69
Metabolic blood test | Before the trail and at the end of cycle 4.
  Number of Participants with abnormal liver function, renal function, blood lipid, blood glucose, blood pressure and other metabolic indicators.
Adverse reactions | From the beginning to 14 days after the end of cycle 4 (each cycle is 28 days).
  It refers to the harmful reaction that has nothing to do with the purpose of treatment in the process of using drugs to prevent, diagnose or treat diseases according to the normal usage and dosage.

CONTACTS AND LOCATIONS:
Overall Officials: naiping wang, Chief physician, Study Director — Dongguan Hospital of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: Yes
The results were published within 6 months after the completion of the test.
Supporting Information: CSR
Time Frame: The results were published within 6 months after the completion of the test.
URL: http://www.dg-tcm.com/